CLINICAL TRIAL: NCT04024462
Title: A Phase III, Randomized, Multicenter, Open-Label, Two-Arm Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Subcutaneous Administration of the Fixed-Dose Combination of Pertuzumab and Trastuzumab in Combination With Chemotherapy in Chinese Patients With HER2-Positive Early Breast Cancer
Brief Title: A Two-Arm Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Subcutaneous Administration of the Fixed-Dose Combination of Pertuzumab and Trastuzumab in Combination With Chemotherapy in Chinese Participants With HER2-Positive Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO41137
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Early Breast Cancer
MeSH Terms: interventions — pertuzumab; Trastuzumab; Doxorubicin; Cyclophosphamide; Docetaxel; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy (Active Comparator): Participants will receive 8 cycles of neoadjuvant chemotherapy: 4 cycles of doxorubicin plus cyclophosphamide (AC) once every 3 weeks (Q3W) followed by docetaxel Q3W for 4 cycles. Pertuzumab and trastuzumab will be given intravenously (IV) for 4 cycles Q3W concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants will undergo surgery. Thereafter, participants will receive an additional 14 cycles of pertuzumab IV and trastuzumab IV for a total of 18 cycles.
  Interventions: Drug: Pertuzumab IV; Drug: Trastuzumab IV; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Procedure: Surgery; Radiation: Post-Operative Radiotherapy; Drug: Hormone Therapy
- Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy (Experimental): Participants will receive 8 cycles of neoadjuvant chemotherapy: 4 cycles of AC Q3W followed by docetaxel Q3W for 4 cycles. The pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) will be given subcutaneously (SC) for 4 cycles (Q3W) concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants will undergo surgery. Thereafter, participants will receive an additional 14 cycles of the PH FDC SC for a total of 18 cycles.
  Interventions: Drug: Pertuzumab and Trastuzumab FDC SC; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Procedure: Surgery; Radiation: Post-Operative Radiotherapy; Drug: Hormone Therapy

INTERVENTIONS:
Drug: Pertuzumab IV — Pertuzumab will be administered as a fixed non-weight-based loading dose of 840-milligrams (mg) IV and then a 420-mg IV maintenance dose Q3W.
  Other Names: Perjeta; RO4368451
  Arms: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy
Drug: Trastuzumab IV — Trastuzumab will be administered as an 8-milligram per kilogram of body weight (mg/kg) IV loading dose and then 6 mg/kg IV maintenance dose Q3W.
  Other Names: Herceptin; RO0452317
  Arms: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy
Drug: Pertuzumab and Trastuzumab FDC SC — The pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) will be administered SC at a fixed non-weight-based dose. A loading dose of 1200 mg SC pertuzumab and 600 mg SC trastuzumab is then followed by a maintenance dose of 600 mg SC pertuzumab and 600 mg SC trastuzumab Q3W.
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; PHESGO™; PH FDC SC; RG6264; RO7198574
  Arms: Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Drug: Doxorubicin — Doxorubicin 60 milligrams per meter squared of body surface area (mg/m^2) will be administered IV on Day 1 of each cycle of treatment (as part of AC Q3W) for Cycles 1-4.
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m^2 will be administered IV on Day 1 of each cycle of treatment (as part of AC Q3W) for Cycles 1-4.
Drug: Docetaxel — Docetaxel 75 mg/m^2 will be administered IV on Day 1 of Cycle 5. At the investigator's discretion the dose may be escalated to 100 mg/m^2 IV for Cycles 6-8 (Q3W) provided no dose-limiting toxicity occurs.
Procedure: Surgery — Participants in both cohorts are scheduled to undergo surgery after 8 cycles of neoadjuvant therapy. Participants may undergo breast-conserving surgery or mastectomy according to routine clinical practice.
Radiation: Post-Operative Radiotherapy — If indicated, radiotherapy is given after chemotherapy and surgery, during adjuvant HER2-targeted therapy and hormone therapy (for hormone-receptor positive disease).
Drug: Hormone Therapy — For hormone receptor positive breast cancer, tamoxifen or aromatase inhibitors will be allowed as adjuvant hormone therapy for postmenopausal participants and with ovarian suppression or ablation for premenopausal participants in countries where it has been registered for this indication. Its use must be consistent with the registered label. Hormone therapy is given after chemotherapy and surgery during adjuvant HER2-targeted therapy.

SUMMARY:
This study will evaluate the pharmacokinetics, efficacy, and safety of the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) as compared with those of the pertuzumab intravenous (IV) and trastuzumab IV formulations in Chinese participants with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) Performance Status greater or equal to (≤)1
* Stage II-IIIC (T2-T4 plus any N, or any T plus N1-3, M0), locally advanced, inflammatory, or early-stage, unilateral, and histologically confirmed invasive breast cancer
* Primary tumor greater than (>)2 centimeters (cm) in diameter, or node-positive disease (clinically or on imaging, and node positivity confirmed with cytology and/or histopathology)
* Human Epidermal Growth Factor Receptor 2 (HER2)-positive breast cancer confirmed by a central laboratory prior to study enrollment. HER2-positive status will be determined based on pretreatment breast biopsy material and defined as 3+ by immunohistochemistry (IHC) and/or positive by HER2 amplification by in situ hybridization (ISH) with a ratio of ≥2 for the number of HER2 gene copies to the number of signals for chromosome 17 copies
* Hormone receptor status of the primary tumor, centrally confirmed
* Patient agreement to undergo mastectomy or breast conserving surgery after neoadjuvant therapy
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue for central confirmation of HER2, hormone receptor status, and PIK3CA mutational analyses
* Baseline left ventricular ejection fraction (LVEF) ≥55% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* For women of childbearing potential (WOCBP) who are sexually active: agreement to remain abstinent (refrain from heterosexual intercourse) or use one highly effective non-hormonal contraceptive method with a failure rate of less than (<)1% per year, or two effective non-hormonal contraceptive methods during the treatment period and for 7 months after the last dose of HER2-targeted therapy, and agreement to refrain from donating eggs during this same period
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom in combination with a spermicidal foam, gel, film, cream, or suppository, and agreement to refrain from donating sperm, as specified in the protocol
* A negative serum pregnancy test must be available prior to randomization for WOCBP (premenopausal women and women <12 months after the onset of menopause), unless they have undergone surgical sterilization (removal of ovaries and/or uterus)
* No major surgical procedure unrelated to breast cancer within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment

Exclusion Criteria:

* Stage IV (metastatic) breast cancer
* History of invasive breast cancer
* History of concurrent or previously treated non-breast malignancies except for appropriately treated 1) non-melanoma skin cancer and/or 2) in situ carcinomas, including cervix, colon, and skin
* Have received any previous systemic therapy (including chemotherapy, immunotherapy, HER2-targeted agents, endocrine therapy [selective estrogen receptor modulators, aromatase inhibitors], and antitumor vaccines) for treatment or prevention of breast cancer, or radiation therapy for treatment of cancer
* Have a past history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) if they have received any systemic therapy for its treatment or radiation therapy to the ipsilateral breast
* High-risk for breast cancer and have received chemopreventative drugs in the past
* Multicentric (multiple tumors involving more than one quadrant) breast cancer, unless all tumors are HER2-positive
* Bilateral breast cancer
* Have undergone an excisional biopsy of primary tumor and/or axillary lymph nodes
* Axillary lymph node dissection (ALND) prior to initiation of neoadjuvant therapy
* Sentinel lymph node biopsy (SLNB) prior to neoadjuvant therapy
* Treatment with any investigational drug within 28 days prior to randomization
* Serious cardiac illness or medical conditions
* Inadequate bone marrow function
* Impaired liver function
* Inadequate renal function with serum creatinine >1.5X upper limit of normal (ULN)
* Current severe, uncontrolled systemic disease that may interfere with planned treatment (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound-healing disorders)
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 7 months after the last dose of HER2-targeted therapy
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Known active liver disease, for example, active viral hepatitis infection (i.e., hepatitis B or hepatitis C), autoimmune hepatic disorders, or sclerosing cholangitis
* Concurrent, serious, uncontrolled infections, or known infection with HIV
* Known hypersensitivity to study drugs, excipients, and/or murine proteins
* Current chronic daily treatment with corticosteroids (dose >10 milligrams [mg] methylprednisolone or equivalent excluding inhaled steroids)
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, colon, skin, and/or non-melanoma skin carcinoma
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe LVSD, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2026-01-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- China (18):
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Hebei Medical University Fourth Hospital, Shijiazhuang
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 18 investigational sites in China.
Pre-assignment Details: Participants with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer, who were candidates for preoperative neoadjuvant treatment in the clinical practice, were enrolled in the study.
Groups:
- Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy: Participants received 8 cycles of neoadjuvant chemotherapy: 4 cycles of doxorubicin plus cyclophosphamide (AC) once every 3 weeks (Q3W) followed by docetaxel Q3W for 4 cycles. Pertuzumab and trastuzumab were given intravenously (IV) for 4 cycles Q3W concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants underwent surgery. Thereafter, participants received an additional 14 cycles of pertuzumab IV and trastuzumab IV for a total of 18 cycles.
- Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy: Participants received 8 cycles of neoadjuvant chemotherapy: 4 cycles of AC Q3W followed by docetaxel Q3W for 4 cycles. The pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) were given subcutaneously (SC) for 4 cycles (Q3W) concurrently with the taxane component of chemotherapy. After completing their neoadjuvant therapy, participants underwent surgery. Thereafter, participants received an additional 14 cycles of the PH FDC SC for a total of 18 cycles.
Period: Overall Study
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Started (Intent-to-Treat (ITT) Population) | 101 | 99
Completed Neoadjuvant Treatment (24 Weeks) | 96 | 95
Completed Surgery (<9 Weeks) | 94 | 93
Started Adjuvant Treatment | 89 | 89
Completed Adjuvant Treatment (42 Weeks) | 12 | 14
Started Follow-Up (≥3 Years) (Participants who completed treatment or prematurely withdrew from treatment entered the follow-up phase.) | 23 | 20
Completed | 0 | 0
Not Completed | 101 | 99
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Progressive Disease | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Ongoing in the Study | 94 | 89

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.17 (10.55) | 50.42 (10.01) | 50.80 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 99 | 200
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 99 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 101 | 99 | 200
Randomization Stratification Factors: Hormone Receptor Status [Count of Participants; unit: Participants] — Hormone receptor status was based on central assessment of participant samples for estrogen receptor (ER) and progesterone receptor (PgR) negativity or positivity.
  Participants
    ER Negative and PgR Negative | 51 | 51 | 102
    ER Positive and PgR Positive | 50 | 48 | 98
Randomization Stratification Factors: Clinical Stage at Presentation [Count of Participants; unit: Participants] — Breast cancer stages range from 0 to IV with IV being the most advanced stage, which is considered a worse outcome. Stages II and III are both invasive breast cancer stages and are subdivided into IIA, IIB, IIIA, IIIB and IIIC based on tumor size, presence and number of metastases in regional lymph nodes and presence of distant metastases. Participants enrolling in this study were categorized into stages II-IIIA and IIIB-IIIC with IIIC being considered the worst stage.
  Participants
    Stage II-IIIA | 70 | 70 | 140
    Stage IIIB-IIIC | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Serum Trough Concentration (Ctrough) of Pertuzumab During Cycle 7 (Pre-Dose Cycle 8)
Description: The observed pertuzumab trough serum concentration (Ctrough) at Cycle 7 was assessed following 3 cycles of pertuzumab IV and trastuzumab IV or the fixed-dose combination (FDC) of pertuzumab and trastuzumab SC. The Per Protocol Pharmacokinetics (PK) analysis population includes all enrolled participants who adhered to the protocol. Exclusions from the Per Protocol PK analysis population were made for the following reasons: participants were missing the Ctrough pre-dose Cycle 8 PK sample, participants with a Ctrough sample collected with at least 2 days deviation from the planned date on Day 21 (i.e., before Day 19 or after Day 23), participants given a dose amount that deviated from the planned dose by >20% within 3 cycles (from Cycle 5), participants with a dose delay of more than 7 days, a Cycle 7 subcutaneous injection site other than thigh was used, if the Cycle 8 IV pre-dose and post-dose PK samples were switched, and an assay error impacting Ctrough measurement.
Time Frame: Pre-dose at Cycle 8 (one cycle is 21 days)
Population: Pertuzumab Per Protocol PK Population: includes only participants who adhered to the pre-specified criteria for the schedule of pharmacokinetic assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 89 | 89
micrograms per millilitre (μg/mL) | 69.9 (30.8) | 74.6 (30.5)
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; The null hypothesis was that the pertuzumab Arm B SC dose is inferior to the pertuzumab Arm A IV dose (i.e., the CtroughSC/CtroughIV geometric mean ratio of the SC dose of pertuzumab relative to the IV dose is not greater than 0.8); Test type: Non-Inferiority — The null hypothesis could be rejected and non-inferiority concluded if the lower bound of the 90% confidence interval of the geometric mean ratio was ≥0.8; Geometric Mean Ratio = 1.07, 90% CI 2-sided [0.99 to 1.15] — The CtroughSC/CtroughIV geometric mean ratio was calculated as the SC dose of pertuzumab (Arm B) relative to the pertuzumab IV dose (Arm A)

2. Primary Outcome: Serum Ctrough of Trastuzumab During Cycle 7 (Pre-Dose Cycle 8)
Description: The observed trastuzumab trough serum concentration (Ctrough) at Cycle 7 was assessed following 3 cycles of pertuzumab IV and trastuzumab IV or the fixed-dose combination (FDC) of pertuzumab and trastuzumab SC. The Per Protocol Pharmacokinetics (PK) analysis population includes all enrolled participants who adhered to the protocol. Exclusions from the Per Protocol PK analysis population were made for the following reasons: participants were missing the Ctrough pre-dose Cycle 8 PK sample, participants with a Ctrough sample collected with at least 2 days deviation from the planned date on Day 21 (i.e., before Day 19 or after Day 23), participants given a dose amount that deviated from the planned dose by >20% within 3 cycles (from Cycle 5), participants with a dose delay of more than 7 days, a Cycle 7 subcutaneous injection site other than thigh was used, if the Cycle 8 IV pre-dose and post-dose PK samples were switched, and an assay error impacting Ctrough measurement.
Time Frame: Pre-dose at Cycle 8 (one cycle is 21 days)
Population: Trastuzumab Per Protocol PK Population: includes only participants who adhered to the pre-specified criteria for the schedule of pharmacokinetic assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milllilitre (μg/mL)
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 89 | 89
micrograms per milllilitre (μg/mL) | 33.6 (28.8) | 52.1 (32.5)
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; The null hypothesis was that the trastuzumab Arm B SC dose is inferior to the Arm A trastuzumab IV dose (i.e., the CtroughSC/CtroughIV geometric mean ratio of the SC dose of trastuzumab relative to the IV dose is not greater than 0.8); Test type: Non-Inferiority — The null hypothesis could be rejected and non-inferiority concluded if the lower bound of the 90% confidence interval of the geometric mean ratio was ≥0.8. Non-inferiority was tested in hierarchical order after the primary outcome measure, to adjust for multiple statistical testing and control the type I error at one sided 5% significance level; Geometric Mean Ratio = 1.55, 90% CI 2-sided [1.44 to 1.67] — The CtroughSC/CtroughIV geometric mean ratio was calculated as the SC dose of trastuzumab (Arm B) relative to the trastuzumab IV dose (Arm A)

3. Secondary Outcome: Percentage of Participants With Total Pathological Complete Response (tpCR), According to Local Pathologist Assessment
Description: Total pathological complete response (tpCR) was defined as eradication of invasive disease in the breast and axilla; that is, ypT0/is ypN0, according to the local pathologists' assessment. Pathologic response to therapy was determined at the time of surgery. The tpCR rate is the percentage of participants in the ITT population who achieved a tpCR. Participants with missing data for tpCR (i.e., do not undergo surgery or have an invalid pCR assessment) were included in the analysis and classified as non-responders. Rates of tpCR were calculated in each treatment arm and were assessed using the difference between the Arm B: Pertuzumab and Trastuzumab FDC SC and the Arm A: Pertuzumab IV and Trastuzumab IV tpCR rates and corresponding 95% Clopper-Pearson confidence intervals (CIs). The difference between the tpCR rates along with corresponding 95% Hauck-Anderson CIs were calculated.
Time Frame: Following completion of surgery (up to 33 weeks)
Population: ITT Population: includes all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
Number analyzed (Participants) | 101 | 99
percentage of participants | 56.4 [46.20 to 66.28] | 55.6 [45.22 to 65.55]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy vs Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy; Test type: Other — Descriptive analysis only. tpCR was analyzed outside of a hypothesis-testing framework and according to the methodology outlined in the outcome measure description; Difference in tpCR Rate = -0.88, 95% CI 2-sided [-15.21 to 13.45] — Difference in tpCR rate was calculated as Arm B: PH FDC SC minus Arm A: P+H IV

4. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to Invasive Disease-Free Survival (iDFS; Excluding Second Primary Non-Breast Cancer [SPNBC]) Criteria
Description: iDFS (excluding SPNBC) is defined as the time from the first date of no disease (i.e., the date of primary surgery) to the first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence; ipsilateral local-regional invasive breast cancer reccurrence; distant recurrence; contralateral invasive breast cancer; or death attributable to any cause. Ipsilateral or contralateral in situ disease and SPNBC (including in situ carcinomas and non-melanoma skin cancers) will not be counted as progressive disease or relapse.
Time Frame: From date of surgery to iDFS (excluding SPNBC) event (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

5. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to iDFS (Including SPNBC) Criteria
Description: iDFS including SPNBC is defined in the same way as iDFS but including SPNBC as an event (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Time Frame: From date of surgery to iDFS (including SPNBC) event (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

6. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to Event-Free Survival (EFS; Excluding SPNBC) Criteria
Description: EFS (excluding SPNBC) is defined as the time from enrollment to the first occurrence of one of the following events: breast cancer progression; breast cancer recurrence; or death from any cause. Ipsilateral or contralateral in situ disease and SPNBC (including in situ carcinomas and non-melanoma skin cancers) will not be counted as progressive disease or relapse.
Time Frame: From baseline to EFS (excluding SPNBC) event (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

7. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to EFS (Including SPNBC) Criteria
Description: EFS including SPNBC is defined in the same way as EFS, but including SPNBC as an event (with the exception of non-melanoma skin cancers and in situ carcinoma of any site).
Time Frame: From baseline to EFS (including SPNBC) event (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

8. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Are Event-Free According to Distant Recurrence-Free Interval (DRFI) Criteria
Description: DRFI is defined as the time between randomization and the date of distant breast cancer recurrence.
Time Frame: From baseline to DFRI event (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

9. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants in Overall Survival
Time Frame: From baseline to death from any cause (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

10. Secondary Outcome: Number of Participants With at Least One Adverse Event by Severity, Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4 (NCI CTCAE v4)
Time Frame: From baseline until study completion (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

11. Secondary Outcome: Number of Participants With a Primary Cardiac Event
Description: A primary cardiac event is defined as either a symptomatic ejection fraction decrease (heart failure) of New York Heart Association (NYHA) Class III/IV and a drop in left ventricular ejection fraction (LVEF) of at least 10-percentage points from baseline and to below 50%, or a definite or probable cardiac death. NYHA Class III is defined as: marked limitation of physical activity; comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. NYHA Class IV is defined as: Inability to carry on any physical activity without discomfort; symptoms of cardiac insufficiency at rest; if any physical activity is undertaken, discomfort is increased. Definite cardiac death is defined as death due to heart failure, myocardial infarction, or documented primary arrhythmia. Probable cardiac death is defined as sudden unexpected death within 24 hours of a definite or probable cardiac event (e.g., syncope, cardiac arrest, chest pain, etc.) without documented etiology.
Time Frame: From baseline until study completion (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

12. Secondary Outcome: Number of Participants With a Secondary Cardiac Event, Defined as an Asymptomatic or Mildly Symptomatic Left Ventricular Systolic Dysfunction (LVSD) of NYHA Class II
Description: An LVSD ("Ejection fraction decreased") of NYHA Class II is defined as a left ventricular ejection fraction (LVEF) decrease of ≥10-percentage points below the baseline measurement to an absolute LVEF value of <50%, confirmed by a second LVEF assessment within approximately 3 weeks also showing a documented drop.
Time Frame: From baseline until study completion (up to 5.5 years)
Reporting Status: Not Posted, anticipated posting 2027-02

ADVERSE EVENTS:
Time Frame: From baseline until the primary completion date (up to approximately 1 year, 10 months)
Description: Adverse events (AEs) were analyzed for the safety analysis population, which included all participants who received at least one dose of study medication, according to the treatment actually received. One participant randomized to Arm A (IV) mistakenly received 1 SC injection of pertuzumab and trastuzumab FDC SC and was counted in Arm B (SC) for safety; total number analyzed in Arm A: 101-1=100, Arm B: 99+1=100. AEs are still being collected and will be updated within 1 year of study completion.
Arm/Group | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/100
Serious Adverse Events (participants affected / at risk) | 19/100 | 18/100
Other Adverse Events (participants affected / at risk) | 96/100 | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy (N=100) | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN FLAP NECROSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (3) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 (3) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FIBROADENOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pertuzumab IV + Trastuzumab IV + Chemotherapy (N=100) | Arm B: Pertuzumab and Trastuzumab FDC SC + Chemotherapy (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 63 (168) | 65 (156)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4) | 7 (8)
LEUKOPENIA (Blood and lymphatic system disorders) | 25 (123) | 17 (103)
NEUTROPENIA (Blood and lymphatic system disorders) | 9 (63) | 9 (50)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 (13) | 7 (9)
CONSTIPATION (Gastrointestinal disorders) | 10 (16) | 12 (23)
DIARRHOEA (Gastrointestinal disorders) | 39 (93) | 27 (53)
MOUTH ULCERATION (Gastrointestinal disorders) | 11 (16) | 14 (23)
NAUSEA (Gastrointestinal disorders) | 48 (99) | 45 (97)
STOMATITIS (Gastrointestinal disorders) | 7 (7) | 6 (11)
TOOTHACHE (Gastrointestinal disorders) | 3 (4) | 6 (12)
VOMITING (Gastrointestinal disorders) | 42 (80) | 46 (91)
INFLUENZA LIKE ILLNESS (General disorders) | 5 (6) | 6 (6)
MALAISE (General disorders) | 15 (28) | 12 (26)
PYREXIA (General disorders) | 15 (19) | 11 (22)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 3 (4)
URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 6 (7)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 10 (14) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 39 (76) | 46 (71)
ALPHA HYDROXYBUTYRATE DEHYDROGENASE INCREASED (Investigations) | 5 (11) | 6 (11)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 39 (76) | 38 (55)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 9 (13) | 12 (16)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 5 (6)
BLOOD CREATININE INCREASED (Investigations) | 2 (5) | 7 (12)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 9 (20) | 8 (15)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7 (10) | 8 (10)
LYMPHOCYTE COUNT DECREASED (Investigations) | 13 (25) | 14 (26)
NEUTROPHIL COUNT DECREASED (Investigations) | 59 (166) | 60 (190)
PLATELET COUNT DECREASED (Investigations) | 18 (51) | 21 (40)
WEIGHT DECREASED (Investigations) | 8 (9) | 8 (8)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 46 (169) | 56 (208)
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 (33) | 11 (29)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 (4) | 9 (11)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 9 (9) | 10 (18)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 12 (14) | 18 (43)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 10 (18) | 11 (20)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 13 (21) | 13 (30)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (6) | 6 (8)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 8 (11) | 4 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (10)
DIZZINESS (Nervous system disorders) | 8 (12) | 4 (7)
HEADACHE (Nervous system disorders) | 5 (7) | 2 (2)
HYPOAESTHESIA (Nervous system disorders) | 6 (9) | 8 (10)
INSOMNIA (Psychiatric disorders) | 2 (2) | 11 (14)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 13 (14)
ALOPECIA (Skin and subcutaneous tissue disorders) | 58 (58) | 66 (66)
RASH (Skin and subcutaneous tissue disorders) | 13 (20) | 15 (27)
HYPERTENSION (Vascular disorders) | 3 (4) | 5 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT04024462/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04024462/SAP_001.pdf